CLINICAL TRIAL: NCT03076710
Title: Two-Stage, Pilot, Prospective, Observational Study of Post-Operative Pain Management Following Spine Surgery
Brief Title: Post-Operative Pain Management Following Spine Surgery
Acronym: EXPAREL
Status: Withdrawn | Type: Observational
Why Stopped: No participants were identified per inclusion/exclusion criteria
Sponsor: University of Miami (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Steven Vanni, Associate Professor, University of Miami
Other Study IDs: 20140496
Record Dates: First submitted 2017-02-24; First posted 2017-03-10 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Pain Management; Analgesia; Anesthetic
Keywords: spine surgery; post-operative pain; patient controlled analgesia; Exparel®; bupivacaine
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Opioids delivered through PCA: PCA devices used to deliver opioids
  Interventions: Drug: Opioids delivered through PCA
- EXPAREL® infiltration: EXPAREL® infiltration at the site of surgery and nurse-administered opioid as needed
  Interventions: Drug: EXPAREL® infiltration

INTERVENTIONS:
Drug: Opioids delivered through PCA — IV up to 1 mg. morphine every 10 minutes on request and oral opioids up to 2 tablets of Percocet every 4 hours
  Groups: Opioids delivered through PCA
Drug: EXPAREL® infiltration — 22 gauge / 3.5" needle, into dermal/fascial/muscular/subcutaneous layers and up to 4mg IV morphine every 60 minutes on request and standardized oral opioids on request
  Other Names: Bupivacaine; Marcaine
  Groups: EXPAREL® infiltration

SUMMARY:
The primary objective of this pilot study is to assess the feasibility of comparing two standardized approaches to manage post-operative pain following spine surgery: one approach using Patient Controlled Analgesia (PCA) devices to deliver opioid analgesics, and the other approach using EXPAREL® infiltration at the site of surgery and nurse-administered opioid analgesics.

DETAILED DESCRIPTION:
The study will assess the feasibility of the methods proposed, including recruitment, eligibility, standardization of both post-operative pain management approaches, and assessment of clinical, hospital efficiency, medication use, health services use, and economic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Ability to speak, read, and write in English or Spanish
* Primary indication is low back pain, radiculopathy, disc degeneration, disc herniation, foraminal stenosis, or mild 1-level spondylolisthesis or deformity
* Scheduled to undergo primary, single level, lumbar fusion surgical procedure at the study center in the next 30 days
* Willing to provide informed consent, participate in study, and comply with study protocol

Exclusion Criteria:

* Body mass index >35
* Pregnant or contemplating pregnancy prior to surgery
* Current or previous psychiatric, behavioral, or emotional disorder that may interfere with postsurgical pain, analgesia, or opioid use according to treating surgeon
* Prior treatment for alcohol, recreational drug, or opioid abuse
* Chronic inflammatory conditions (e.g. Crohn's, lupus, rheumatoid arthritis)
* Chronic neurologic conditions (e.g. multiple sclerosis, Parkinson's)
* Serious spinal conditions (e.g. cauda equina syndrome, infection, tumor, fracture)
* Hypersensitivity or allergy to local anesthetics
* Previous surgery in lumbar spine (i.e. other than microdiscectomy);
* Continuous (e.g. daily) opioid consumption for more than 30 days prior to surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary, single level, lumbar fusion surgical procedures.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Pain severity at the site of surgery | 4 hours post surgery
  Numerical Rating Scale 0 (no pain) to 10 (worst pain imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Vanni, DO, DC, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No